CLINICAL TRIAL: NCT04532372
Title: A Phase 1/2 Trial of Leflunomide for the Treatment of Severe COVID-19 in Patients With a Concurrent Malignancy
Brief Title: Leflunomide for the Treatment of Severe COVID-19 in Patients With a Concurrent Malignancy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20291; NCI-2020-05746 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20291 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Symptomatic COVID-19 Infection Laboratory-Confirmed
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Leflunomide

STUDY DESIGN:
Intervention Model Description: Phase I single-arm dose-escalation design followed by a phase II randomized two-arm design
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I (leflunomide, SOC) (Experimental): Patients receive leflunomide PO QD on days 1-14. Patients may receive SOC drugs in addition to leflunomide.
  Interventions: Other: Best Practice; Drug: Leflunomide
- Phase II Arm I (leflunomide, SOC) (Experimental): Patients receive leflunomide PO QD on days 1-14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive SOC.
  Interventions: Other: Best Practice; Drug: Leflunomide; Drug: Placebo Administration
- Phase II Arm II (placebo, SOC) (Placebo Comparator): Patients receive placebo PO QD on days 1-14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive SOC.
  Interventions: Other: Best Practice; Drug: Placebo Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care drugs
  Other Names: standard of care; standard therapy
Drug: Leflunomide — Given PO
  Other Names: Arava; SU101
  Arms: Phase I (leflunomide, SOC); Phase II Arm I (leflunomide, SOC)
Drug: Placebo Administration — Given PO
  Arms: Phase II Arm I (leflunomide, SOC); Phase II Arm II (placebo, SOC)

SUMMARY:
This phase I/II trial investigates the best dose and side effects of leflunomide and how well it works in treating patients with COVID-19 and a past or present cancer. Leflunomide has been used since the 1990s as a treatment for rheumatoid arthritis. Experiments done with human cells that were given severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus causing COVID-19, showed that leflunomide was able to reduce the ability of the virus to make copies of itself. The coronavirus uses ribonucleic acid (RNA), a very long molecule that contains genetic information that is like a blueprint for making more copies of itself. Leflunomide inhibits the formation of RNA. The information gained from this study may help researchers to learn whether leflunomide is safe for use in treating patients with COVID-19, and whether it is potentially effective against the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and tolerability of leflunomide when combined with coronavirus disease 2019 (COVID-19) standard of care (SOC) by evaluation of toxicities including: type, frequency, severity, attribution and duration. (Phase 1) II. Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of leflunomide when given in combination with SOC. (Phase 1) III. Evaluate the clinical activity of leflunomide plus SOC (Arm 1) and placebo plus SOC (Arm 2) on the basis of clinical improvement (response) rate in each treatment arm, as assessed by a 7-point ordinal scale. (Phase 2/Pilot) IV. Evaluate the safety and tolerability of leflunomide plus SOC (Arm 1) and placebo plus SOC (Arm2). (Phase 2/Pilot)

SECONDARY OBJECTIVES I. Evaluate the clinical activity of leflunomide when combined with SOC on the basis of clinical improvement (response) rate. (Phase 1)

II. Estimate the following (Phase 1 and Phase 2):

IIa.Time to clinical improvement (days). IIb. Time to peripheral capillary oxygen saturation (SpO2) > 93% on room air (days).

IIc. Time to first negative SARS-CoV-2 polymerase chain reaction (PCR) (days). IId. Duration of oxygen therapy (days). IIe. Duration of hospitalization (days). IIf. Duration of mechanical ventilation. IIg. All cause mortality at day 28. III. Measure trough plasma concentrations of the active metabolite teriflunomide on days 1 through 14, day 21, and day 28, and evaluate relationships between teriflunomide levels and pharmacodynamic biomarkers (e.g., viral load, cytokines), response, safety, and concomitant medications. (Phase 1 and Phase 2)

EXPLORATORY OBJECTIVES

I. Investigate inflammatory response by measuring changes before and after leflunomide treatment in:

Ia. Circulating cytokines (e.g., IL-6, IL-8, TNF-alpha, IL-12, interferons [IFNs] and granulocyte-macrophage colony-stimulating factor ([GM-CSF]).

Ib. Immune effector cell phenotype associated with monocyte, T cell, and natural killer (NK) cell activation.

II. Assess the kinetics of viral replication through serial measurements of viral load by nasopharyngeal swab and tracheal aspirates (if on ventilator and can be safely obtained).

OUTLINE: This is a phase I dose-escalation study, followed by a phase II study.

PHASE I: Patients receive leflunomide orally (PO) once daily (QD) on days 1-14. Patients may receive SOC drugs in addition to leflunomide.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I (LEFLUNOMIDE + SOC): Patients receive leflunomide PO QD on days 1-14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive SOC.

ARM II (PLACEBO + SOC): Patients receive placebo PO QD on days 1-14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive SOC.

After completion of study treatment, patients are followed up for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative. Assent, when appropriate, will be obtained per institutional guidelines. Cognitively impaired subjects may enroll in the phase 2 portion if adequate psychosocial support is provided
* SARS-CoV-2 infection confirmed by a PCR-based test within 4 days prior to enrollment
* COVID-19 disease baseline severity of Severe according to FDA guidance, as defined by:

  * Symptoms suggestive of severe systemic illness with COVID-19, which could include any symptom of fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, or shortness of breath at rest, or respiratory distress
  * Clinical signs indicative of severe systemic illness with COVID-19, such as respiratory rate >= 30 per minute, heart rate >= 125 per minute, SpO2 =< 93% on room air at sea level or partial pressure of oxygen (PaO2)/the fraction of inspired oxygen (FiO2) < 300
* Active cancer requiring systemic treatment within the last 2 years. Subjects should not have received the following therapies for their malignancy within the indicated time frames:

  * Local radiation therapy within 2 weeks prior to enrollment. If the involved field is small (single nodal area), 7 days prior to enrollment is allowed
  * Chemotherapy within 2 weeks prior to enrollment
  * Major surgery within 2 weeks prior to treatment
  * Autologous hematopoietic stem cell infusion within 12 weeks prior to enrollment
  * Antibody therapy, chimeric antigen receptor (CAR) T cells, or other biologic therapies within 12 weeks prior to enrollment
  * Allogeneic hematopoietic stem cell infusion within 16 weeks prior to enrollment These time frames should be considered the minimum allowed interval and may be longer per the judgment of the investigator
* Adverse events related to prior cancer therapy must have recovered to =< grade 1 or to baseline
* Subjects must be able to forgo systemic cancer therapy for ~39 days (14 days treatment/placebo + 14 days monitoring + ~ 11 days cholestyramine)
* Absolute neutrophil cunt (ANC) >= 500/mm^3 (to be performed within 4 days prior to day 1 of protocol therapy unless otherwise stated)
* Platelets >= 25,000/mm^3 (to be performed within 4 days prior to day 1 of protocol therapy unless otherwise stated)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (unless has Gilbert's disease) (to be performed within 4 days prior to day 1 of protocol therapy unless otherwise stated)
* Aspartate aminotransferase (AST) =< 2 x ULN (to be performed within 4 days prior to day 1 of protocol therapy unless otherwise stated)
* Alanine aminotransferase (ALT) =< 2 x ULN (to be performed within 4 days prior to day 1 of protocol therapy unless otherwise stated)
* Creatinine clearance of >= 60 mL/min per 24-hour urine test or the Cockcroft-Gault formula (to be performed within 4 days prior to day 1 of protocol therapy unless otherwise stated)
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study until teriflunomide levels are verified to be less than 0.02 mg/L (0.02 ug/mL) for patients given leflunomide, or until unblinding occurs for those given placebo. Contraception should also be used for the duration of administration of SOC drugs during this study for the duration recommended in the prescribing information.

  * Childbearing potential is defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Evidence of acute respiratory distress syndrome (ARDS), defined by at least one of the following: endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates > 20 L/min with fraction of delivered oxygen >= 0.5), noninvasive positive pressure ventilation, extracorporeal membrane oxygenation (ECMO), or clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation)
* Shock (defined by systolic blood pressure < 90 mm Hg, or diastolic blood pressure < 60 mm Hg or requiring vasopressors)
* Evidence of multi-organ dysfunction/failure
* Pre-existing acute or chronic liver disease
* Patients with indolent local malignancies or pre-malignant conditions including but not limited to:

  * Smoldering multiple myeloma or monoclonal gammopathy of undetermined significance (MGUS)
  * Basal or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix or breast
  * Incidental histologic finding of prostate cancer (T1a or T1b using the tumor node metastasis [TNM] clinical staging system) or prostate cancer that is curative
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Secondary bacterial, fungal, or viral infections that are not adequately controlled
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* If human immunodeficiency virus (HIV)-positive: CD4+ T cell count < 200
* Positive for tuberculosis antigen (e.g., T-spot test)
* Presence of liver metastasis
* Gastrointestinal (GI) malignancies associated with malabsorption and inability to take cholestyramine
* Steroids, except for low-dose replacement or high-dose for management of acute symptoms such as ARDS
* Any new immunosuppressive medication in the 4 weeks prior to enrollment, excepting agents used for treatment of COVID-19 that may also have immunosuppressive properties
* Medications that are CYP1A2 inducers, CYP2C8 inhibitors, and vitamin K antagonists, if these medications are not approved by the investigator. CYP1A2 inducers, CYP2C8 inhibitors, and vitamin K antagonists that are approved by the investigator are allowed
* Concurrent administration of live vaccines
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeet S Dadwal, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase I (Leflunomide, SOC) | Phase II Arm I (Leflunomide, SOC) | Phase II Arm II (Placebo, SOC)
Started | 2 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to the low accrual rate, the study was terminated after two subjects enrolled in Phase I.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I (Leflunomide, SOC) | Phase II Arm I (Leflunomide, SOC) | Phase II Arm II (Placebo, SOC) | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 71.5 [55 to 88] |  |  | 71.5 [55 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  |  | 2
  Male | 0 |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  | 0
  Not Hispanic or Latino | 2 |  |  | 2
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 1 |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 1 |  |  | 1
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase 1)
Description: MTD were based on the assessment of DLT (Dose Limiting Toxicity) during the 28-day treatment period.
Time Frame: From the initial study treatment (Day 0) to Day 28.
Population: Due to the low accrual rate, the study was terminated after two subjects enrolled in Phase I.
Measure: Number; unit: mg
Arm/Group | Phase I (Leflunomide, SOC)
Number analyzed (Participants) | 2
mg | NA — Per study design, to determine MTD, it needs to have at least five accruals. So, MTD is unable to be determined for this study.

2. Primary Outcome: Clinical Activity (Response)(Phase 2)
Description: Defined as a >= 2-point change in clinical status from day 1 on a 7-point ordinal scale. The ordinal scale is an assessment of the clinical status at a given study day. Each day, the worst (i.e., lowest ordinal) score from the previous day was recorded.
Time Frame: At day 28
Population: Due to the low accrual rate, the study was terminated after two subjects enrolled in Phase I. Therefore, there is no accrual in Phase II.
Arm/Group | Phase II Arm I (Leflunomide, SOC) | Phase II Arm II (Placebo, SOC)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Clinical Activity (Response)
Description: Defined as time from start of treatment to >= 2-point change in clinical status on a 7-point ordinal scale. The ordinal scale is an assessment of the clinical status at a given study day. Each day, the worst (i.e., lowest ordinal) score from the previous day was recorded.
Time Frame: Up to 28 days
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Groups:
- Phase II Arm I (Placebo, SOC): Patients receive leflunomide PO QD on days 1-14. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive SOC.
  Best Practice: Receive standard of care drugs
  Leflunomide: Given PO
  Placebo Administration: Given PO
Arm/Group | Phase I (Leflunomide, SOC) | Phase II Arm I (Placebo, SOC) | Phase II Arm II (Placebo, SOC)
Number analyzed (Participants) | 2 | 0 | 0
days | 9.5 [5 to 14] |  |

4. Secondary Outcome: Overall Survival (Phase 2)
Description: Defined as time from start of treatment to death from any cause
Time Frame: Up to 90 days
Population: as for outcome 2
Arm/Group | Phase II Arm I (Leflunomide, SOC) | Phase II Arm II (Placebo, SOC)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Oxygen Saturation Improvement
Description: Time from start of treatment to peripheral capillary oxygen saturation (SpO2) > 93% on room air.
Time Frame: Up to 90 days
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Phase I (Leflunomide, SOC) | Phase II Arm I (Leflunomide, SOC) | Phase II Arm II (Placebo, SOC)
Number analyzed (Participants) | 2 | 0 | 0
days | 6.5 [1 to 12] |  |

6. Secondary Outcome: Number of Participants Who Were Hospitalized
Description: Indicate the participants who were hospitalized within first 90 days following start of treatment assessed.
Time Frame: Up to 90 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (Leflunomide, SOC) | Phase II Arm I (Leflunomide, SOC) | Phase II Arm II (Placebo, SOC)
Number analyzed (Participants) | 2 | 0 | 0
Participants | 2 |  |

7. Secondary Outcome: Number of Participants Who Were Mechanical Ventilation Required
Description: Indication the participants who were required mechanical ventilation at any time from start of treatment through 90 days post.
Time Frame: Up to 90 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (Leflunomide, SOC) | Phase II Arm I (Leflunomide, SOC) | Phase II Arm II (Placebo, SOC)
Number analyzed (Participants) | 2 | 0 | 0
Participants | 0 |  |

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and assessed from initial treatment to the end of the study, at D1, D2, D3, D4, D5, D6, D7, D8-14, D15-28, D42, D56, D70 and D90. Vital status was assessed from the initial treatment to the end of the study, up to 90 days after the end of the treatment.
Arm/Group | Phase I (Leflunomide, SOC)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (Leflunomide, SOC) (N=2)
ANEMIA (Blood and lymphatic system disorders) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
FEVER (General disorders) | 1 (1)
GENERALIZED EDEMA (General disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (3)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (2)
PLATELET COUNT DECREASED (Investigations) | 2 (3)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 (3)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (2)
OBESITY (Metabolism and nutrition disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
ANOSMIA (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
NOCTURIA (Renal and urinary disorders) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (3)
HYPOTENSION (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT04532372/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT04532372/ICF_001.pdf